CLINICAL TRIAL: NCT06751940
Title: A Multicenter Clinical Study of Personalized Tumor Neoantigen-loaded DC Vaccine Combined with Conventional Second-line Therapy for the Treatment of Colorectal Cancer Progressed After First-line Treatment
Brief Title: Neoantigen-loaded DC Vaccine and Conventional Second-line Therapy for CRC Progressed After First-line Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISL2024312
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Tumor Neoantigen; DC Vaccine; Colorectal Cancer (CRC); Immunotherapy; Second-line Therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combinational treatment of conventional second-line therapy and neoantigen-loaded DC vaccine (Experimental): Participants will receive a conventional second-line therapy and 10 subcutaneous injections of the vaccine within a treatment period of 21 weeks.
  Interventions: Combination Product: Conventional second-line therapy; Drug: Neoantigen-loaded DC vaccine

INTERVENTIONS:
Combination Product: Conventional second-line therapy — Conventional second-line therapy includes chemotherapy, targeted cancer drugs, and/or PD-1 inhibitors.The chemotherapy drugs, dosage and treatment cycle are determined by the subject's attending physician based on the subject's specific conditions. The medication, dosage and treatment cycle of targeted cancer drugs will be determined by the subject's attending physician based on the subject's specific circumstances. The PD-1 inhibitor treatment cycle is 3 weeks, and the drug is administered by intravenous infusion on the first day (D1) of each treatment cycle. The dosage is based on the instructions.
Drug: Neoantigen-loaded DC vaccine — The treatment with personalized tumor neoantigen-loaded DC vaccine is divided into two periods: the primary phase and the boost phase. The primary phase consists of 6 treatments, with the first 3 treatments spaced one week apart and the subsequent 3 treatments spaced two weeks apart. Vaccine will be administrated on the fourth day (D4) of that week. The boost phase consists of 4 treatments, each spaced three weeks apart. Vaccine will be administrated on the fourth day (D4) of that week.

SUMMARY:
In this study, the investigators provide a combined treatment of personalized tumor neoantigen-loaded DC vaccine and conventional second-line therapy to patients with colorectal cancer (CRC) progressed after first-line treatment. The investigators observe the objective response rate (ORR), disease control rate (DCR), adverse event (AE), serious adverse event (SAE), progression-free survival (PFS), and overall survival (OS) , aiming to evaluate the effectiveness and safety of the treatment.

DETAILED DESCRIPTION:
This study is conducted in accordance with the Declaration of Helsinki and the guidelines of the Consolidated Standards of Reporting Trials.

10 patients with CRC progressed after first-line therapy will be recruited in this study. With doctor's assessment, a combined treatment of conventional second-line therapy and personalized tumor neoantigen-loaded DC vaccine treatment plan will be designed for each participant.

Here are the steps for preparing the neoantigen-loaded DC vaccine:

Collecting venous blood samples; Blood PBMC exome sequencing; RNA transcriptome sequencing; Classifying HLA alleles; Performing bioinformatics analysis, finding meaningful mutations and about 20 neoantigen sequences for each patient; Synthesizing neoantigens; Use a blood apheresis device to collect the patient's blood, isolate the PBMC needed to prepare DC cells, and return the remaining blood components to the patient's body (approximately 10^9 cells will be collected);Preparation of the personalized tumor neoantigen-loaded DC vaccine.

Participants will receive a conventional second-line therapy course and 10 subcutaneous injections of the vaccine within a treatment period of 21 weeks. After treatment, participants will be followed in every 6 weeks till the end of the study. Venous blood collection, physical examination, ECOG Performance Status Scale assessment, CT/MRI scan, X-ray examination, laboratory examination, and other necessary examinations are required at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed CRC;
* At least one measurable lesion;
* Aged 18-70, regardless of gender;
* Disease progression after standard first-line therapy, and more than 2 weeks since the end of the last antitumor treatment;
* Expected survival of ≥3 months;
* ECOG performance status of 0-1;
* Female patients of childbearing age must have a negative pregnancy test and be able to take effective contraceptive measures with no plans for pregnancy within six months of the study;
* Able to undergo all screening period laboratory tests as required by the protocol;
* Normal major organ function, such as heart, liver, and kidney;
* Hematologic parameters: neutrophil count ≥1.5×10^9/L, hemoglobin ≥10g/dL, platelet count ≥100×10^9/L, total bilirubin ≤1.5 times the upper limit of normal, AST and ALT ≤2.5 times the upper limit of normal, creatinine and blood urea nitrogen ≤1.5 times the upper limit of normal, activated partial thromboplastin time ≤1.5×ULN, and International Normalized Ratio or prothrombin time ≤1.5×ULN;
* No active hepatitis, AIDS, syphilis, or other infectious diseases;
* Rheumatoid panel: C-reactive protein (CRP) ≤10.0mg/L; Anti-streptolysin O (ASO) <500U; Erythrocyte sedimentation rate ≤15mm/h (men) or 20mm/h (women);
* Thyroid function tests: 0.27mIU/L ≤ Thyroid-stimulating hormone (TSH) ≤ 4.2mIU/L; 3.1pmol/L ≤ Free triiodothyronine (FT3) ≤ 6.8pmol/L; 12pmol/L ≤ Serum free thyroxine (FT4) ≤ 22pmol/L; 1.3nmol/L ≤ Serum total triiodothyronine (TT3) ≤ 3.1nmol/L; 66nmol/L ≤ Serum total thyroxine (TT4) ≤ 181nmol/L;
* Adrenocorticotropic hormone (ACTH): 1.1-17.6pmol/L;
* Ability to understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

Disease-specific exclusion criteria:

* Patients with uncontrollable brain metastases;
* Subjects expected to require any form of antitumor treatment during the study, including maintenance therapy with other drugs, chemotherapy, and/or surgical resection.

Exclusion criteria for medical history and comorbidities:

* Subjects who have required systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent) or other immunosuppressants within 14 days before the first dose. Inhalational or topical corticosteroids are allowed in the absence of active autoimmune diseases;
* Subjects who have been treated with anticancer immunotherapies or other immunostimulatory anticancer drugs (interferons, interleukins, thymosin, immune cell therapy, etc.) within 3 months before the first dose;
* Subjects participating in other clinical trials or whose first dose is less than 4 weeks (or 5 half-lives of the study drug) after the end of the previous clinical trial (last dose);
* Subjects with severe cardiovascular diseases, such as those meeting NYHA Class II or higher criteria, myocardial infarction, or cerebrovascular accidents (cerebral ischemia, symptomatic cerebral embolism, etc.) occurring within 3 months before the first dose, or unstable arrhythmias or unstable angina within 1 month before starting study treatment;
* Subjects with uncontrolled myocardial ischemia or myocardial infarction, poorly controlled arrhythmias are excluded;
* Subjects with hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg) (Note: a stable antihypertensive regimen should be in place within 1 week before the first dose);
* Subjects who have had significant clinically relevant bleeding symptoms or a clear bleeding tendency within 3 months before the first dose, as well as tumors that have invaded major blood vessels or, in the investigator's judgment, are highly likely to invade major blood vessels and cause major bleeding during treatment. Subjects with obvious hemoptysis, coughing up 2.5 mL or more of blood in the month before the first dose;
* Subjects who have experienced arterial/venous thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral embolism), deep vein thrombosis, and pulmonary embolism, within 3 months before screening;
* Subjects with active tuberculosis;
* Subjects who have had a serious infection within 4 weeks before the first dose, including but not limited to infections requiring hospitalization, bacteremia, severe pneumonia, etc.; Subjects with any active infection;
* Subjects preparing for or who have previously undergone tissue/organ transplantation;
* Subjects with uncontrolled epilepsy, central nervous system disorders, or neurological diseases resulting in cognitive impairment;
* Subjects with a history of splenectomy.

Other exclusion criteria:

* Pregnant or breastfeeding women;
* Subjects with a severe history of allergies or atopic constitution;
* Subjects with a history of chronic alcohol or drug abuse within 6 months before enrollment;
* Subjects deemed unsuitable for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 32 weeks
  According to RECIST (version 1.1) criteria, the proportion of subjects experiencing Complete Response (CR) or Partial Response (PR) within the analyzed population. Provide the 95% CI for the Objective Response Rate (ORR).
Disease control rate (DCR) | Through study completion, an average of 32 weeks
  According to RECIST (version 1.1) criteria, the proportion of subjects experiencing Complete Response (CR), Partial Response (PR), or Stable Disease (SD) within the analyzed population. Provide the 95% CI for the Disease Control Rate (DCR).
Drug safety | Through study completion, an average of 32 weeks
  Safety analysis will be based on data from the safety population. It will primarily involve descriptive statistical analysis, with tables describing the adverse events that occurred in this study.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of recruiting until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 66 months
  Progression-Free Survival (PFS) is defined as the time from the first administration of the study drug to disease progression or death. For subjects who have not reported disease progression at the time of analysis, the date of their last disease progression-free check will be used as the censoring date. The median PFS and its 95% CI will be analyzed using the Kaplan-Meier method, and survival curves will be plotted.
Overall Survival (OS) | From date of recruiting until the date of death from any cause, whichever came first, assessed up to 66 months
  Overall Survival (OS) is defined as the time from the first administration of the study drug to death from any cause. For subjects who have not reported death at the time of analysis, the date of their last known survival will be used as the censoring date. The median OS and its 95% CI will be analyzed using the Kaplan-Meier method, and survival curves will be plotted.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Nanchang, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No